CLINICAL TRIAL: NCT03137563
Title: Evaluation of the Acceptability of HPV Self-sampling Among French Women Eligible for Cervical Cancer Screening
Brief Title: Acceptability of HPV-self Sampling
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Dépistages34 (Montpellier - France) (Unknown); Adoc11 (Carcassonne - France) (Unknown); Maison médicale Paul Valéry - Union Languedoc Mutualité - (Montpellier -France) (Unknown)
Responsible Party: Sponsor
Other Study IDs: UF9839
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Cervical Cancer
Keywords: Women; 25-65 years
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women eligible for cervical cancer screening: French women aged 25 to 65 years living in the Department of Hérault or Aude (France), attending one of the 8 centers where the questionnaire will be distributed
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — The questionnaire will be distributed and collected by the same investigator in one of the eight centers involved in the study. The investigator will verify the inclusion criteria and the absence of exclusion criteria.
  Other Names: Distribution of an anonymous questionnaire

SUMMARY:
This trial aimed at evaluating the acceptability of HPV self-sampling among french women eligible for cervical cancer screening (25 - 65 years old) in the region of Occitanie, in the south of France. Acceptability will be evaluated using an anonymous questionnaire and the main outcome of the study will be the response acceptability " yes " or " no " for HPV self-sampling. Secondary outcome will be analysis of socioeconomic determinants for the acceptability of HPV self-sampling.

These data will help to propose new strategies for cervical cancer screening in France, particularly to taget non-attenting populations

DETAILED DESCRIPTION:
Women will be recruted in 8 centers located in 2 departments , Aude and Herault (in the Region of Occitanie in the south of France).The questionnaire will be proposed to the women attending one of these eight centers by an investigator, who will verify the inclusion and exclusion criteria. The same person will collect the filled questionnaire.

The questionnaire is anonymous and is composed of 15 questions evaluating the acceptability of HPV self-sampling and socio-economic determinants.

These questionnaires will be collected and statistical analysis will be performed using appropriate tools.

This study will bring informations on the acceptibility of HPV self sampling among french women eligible for cervical cancer screening in 2 Departements of the South of France. Self-sampling acceptability will be linked to socio-economic determinants.

These data will be important to propose and evaluate new strategies to improve screening coverage, particularly of the context of the organized cervical cancer screening that will take place in France in 2018.

ELIGIBILITY:
Inclusion Criteria:

* Women 25-65 years old
* Living in the Aude or Herault departments
* Informed patient Exclusion criteria
* Virgins
* Previous hysterectomy
* Present or previous cervical pathology
* Patient under guardianship or tutorship

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women attending 8 centers of the Departments of Hearault and Aude : social medical cares, Department of gynecology in the hospitals of Montpellier and Carcassonne ; mid-wifes consultations.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
accept HPV self-sampling for cervical cancer | 1 day
  Response " Yes " or " No " to the question " would you accept HPV self-sampling for cervical cancer screening ?

SECONDARY OUTCOMES:
Socioeconomic determinants of the response | 1 day
  Socioeconomic determinants of the response " yes " or " no " to the question " would you accept HPV self-sampling for cervical cancer screening ?

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BOULLE, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

REFERENCES:
- [Result] Bertucci M, Bonnet E, Satger L, Kreiche A, Chappert JL, Loy-Morel S, Segondy M, Daures JP, Boulle N. Acceptability of vaginal self-sampling with high-risk human papillomavirus testing for cervical cancer screening: a French questionnaire-based study. Women Health. 2021 Jan;61(1):83-94. doi: 10.1080/03630242.2020.1831683. Epub 2020 Oct 26. PMID 33106125